CLINICAL TRIAL: NCT05055024
Title: A 6-Month Multicenter, Open-Labelled Extension of the Clinical Trial NLS-1021 in Narcoleptic Patients With and Without Cataplexy
Brief Title: An Open Label Study of NLS-2 (Mazindol Extended Release) in Subjects With Narcolepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NLS Pharmaceutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLS-1022
Record Dates: First submitted 2021-09-01; First posted 2021-09-23 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Narcolepsy With Cataplexy; Narcolepsy; Narcolepsy Without Cataplexy
MeSH Terms: conditions — Narcolepsy | interventions — Mazindol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NLS-2 (mazindol extended release) (Experimental): NLS-2 (mazindol extended release) administered once a day.
  Interventions: Drug: Mazindol

INTERVENTIONS:
Drug: Mazindol — Drug: NLS-2
  Other Names: NLS-2; mazindol extended release

SUMMARY:
This is a multicenter, open-label extension of the clinical study NLS-1021, evaluating long-term safety, tolerability, pharmacokinetics (PK), and therapeutic response to treatment with NLS-2 in adult subjects with narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

* The subject must complete all Study NLS-1021 study requirements and assessments up to Visit 6;
* The subject is able, in the opinion of the Investigator, to receive NLS-2 for the 24-week Treatment Phase of this study;
* Biological females of childbearing potential must agree to use a medically acceptable double-barrier method of contraception for at least 30 days prior to Day 1 and until completion of the study;
* The subject is able to comply with the open-labelled extension design schedule and other study requirements;
* The subject provides written informed consent for the open-label extension study.

Exclusion Criteria:

* The subject meets any Exclusion Criteria for Study NLS-1021 at Visit 6 of that study;
* The subject receives any investigational drug (other than the COVID-19 vaccine) that is not NLS-2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of NLS-2 in adult subjects with narcolepsy type 1 (NT1) or narcolepsy type 2 (NT2) | 24 weeks
  Summaries of the number and percentage of subjects who experienced Treatment Emergent Adverse Events (TEAEs), TEAEs related to study drug, SAEs, or discontinued study drug or withdrew from the study due to an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Camozzi, MD, Study Director — NLS Pharmaceutics
Locations (22):
- United States (22):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Stanford Sleep Medicine Center, Redwood City, California
  - Pacific Research Network, San Diego, California
  - St. Francis Sleep Allergy and Lung Institute, Clearwater, Florida
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - Ivetmar Medical Group, Miami, Florida
  - The Angel Medical Research Corporation, Miami Lakes, Florida
  - Treken Primary care, Atlanta, Georgia
  - NeuroTrials Research, Atlanta, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - Hawaii Pacific Neuroscience Clinical Research Center, Honolulu, Hawaii
  - The Center For Sleep & Wake Disorders, Chevy Chase, Maryland
  - Sleep and Attention Disorders, Sterling Heights, Michigan
  - Neurology and Sleep Disorders Clinic, Columbia, Missouri
  - Carolinas Sleep Specialists, Concord, North Carolina
  - Superior Clinical Research, LLC, Goldsboro, North Carolina
  - Advanced Respiratory and Sleep Medicine, Huntersville, North Carolina
  - Intrepid Research, Cincinnati, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Bogan Sleep Consultants, Columbia, South Carolina
  - Dharma PA d/b/a Southwest Family Medicine Associates, Dallas, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No